Study Protocol with Statistical Analysis Plan (SAP) and Informed Consent Form (ICF)

**Study Protocol** 

(Pages 2 – 6)

**January 11, 2018** 

#### **Study Protocol**

The study titled "The Effects of a Hippotherapy Simulator in Children with Cerebral Palsy" was approved by the Marmara University Faculty of Medicine Clinical Researches Ethics Committee meeting on 02.09.2016 with approval number: 09.2016.478 (Annex-1).

This study was conducted in "The Private Dilbade Special Education and Rehabilitation Center" between 14.12.2016 and 28.10.2017 with 30 children with spastic Cerebral Palsy (CP) who agreed to participate in the study.

The legal representatives of the children who participated in the study were informed about the aim, duration and the programs to be applied throughout the study. Volunteer Information Form has been signed and approved by the standards deemed appropriate by the Clinical Researches Ethics Committee of Marmara University Faculty of Medicine (This form can be seen on Informed Consent Form (ICF) section). The study was conducted by the Declaration of Helsinki.

#### The hypothesis of the Study

H0: Addition of the exercises performed with Hippotherapy Simulator (HS) device to the Neurodevelopmental Therapy (NDT) based rehabilitation program in children with CP does not contribute positively in improving the efficiency of gross motor functions, lower extremity functions, muscle tone and spasticity, trunk control, sitting and standing balance, walking functions and functional independence.

H1: Addition of the exercises performed with HS device to the NDT based rehabilitation program in children with cerebral palsy contributes positively to improve the efficiency of gross motor functions, lower extremity functions, muscle tone and spasticity, trunk control, sitting and standing balance, walking functions and functional independence.

#### Randomization of the Study Groups

Children with CP who received rehabilitation services in "The Private Dilbade Special Education and Rehabilitation Center" were invited to participate in the study. Two different treatment methods were applied to the children who volunteered to participate and met the participation criteria. Rehabilitation programs based on individual NDT were applied to the children included in the study for eight weeks (first group). In the next eight weeks, the HS

system was applied to the same children in addition to individual NDT based rehabilitation programs (study group).

#### **Inclusion Criteria**

- Having a diagnosis of Spastic CP,
- Children aged between 5 18 years,
- GMFCS level is I, II or III,
- Independent seating,
- Walking with at least 10 meters of independent, orthotic and/or auxiliary device,
- Can understand simple verbal instruction,
- Those with hip adductor muscle spasticity level less than 2 according to MAS,
- Having bilateral passive hip abduction enough to could sit into the hippotherapy simulator device,
- Voluntarily agreed to participate in the study.

#### **Exclusion Criteria**

- Those with hip dislocation,
- Severe contracture or deformity to prevent the study,
- Advanced scoliosis (above 20 degrees),
- Acute uncontrolled acute seizures,
- Uncontrollable severe epileptic attacks,
- Visual and auditory problems,
- Injection of botulinum toxin in the last 6 months patients,
- Underwent surgical operation such as muscle relaxation, tendon extension and selective dorsal rhizotomy in the last 6 months.

#### **Applied Evaluations**

Evaluations were applied three times: before treatment, after individual NDT programs (at the end of the 8th. week), and after NDT + HS application (at the end of the 16th week). All evaluation data were noted to the "Participant Tracking Form" (Annex-2).

Functional levels of participants were evaluated with the "Gross Motor Function Classification System" (GMFSS). Gross motor functions with "Gross Motor Function Measure-

88" (GMFM-88); lower extremity joint range of motion (ROM) with "universal goniometer"; muscle tones and spasticity with "Modified Ashworth Scale" (MAS) and "Myoton®PRO Digital Palpation Device" was evaluated.

"The Trunk Impairment Scale" (TIS) was used to assess the functional strength of the body, its postural control and the nature of the trunk movements. The Pediatric Balance Scale (PBS), an assessment tool adapted from the Berg Balance Scale (BBS), was used to assess children's functional and dynamic balances in daily life activities. Besides, the Pedalo® Sensamove Balance Test device was used to evaluate the dynamic balance of children in sitting and standing positions. The Functional Independence Measure (WeeFIM) for children was used to assess children's functional independence in daily activities. Win-Track (Medicapteurs, France) path and software system was used to evaluate the walking functions (Spatio-temporal parameters) of children.

#### **Treatment Program**

The participants were selected for the rehabilitation program in "The Private Dilbade Special Education and Rehabilitation Center" twice a week for 16 weeks (duration of one session is 45 minutes).

Firstly, children participating in the study were included in the rehabilitation program using only the NDT approach for 16 sessions (8 weeks x 2 days x 45 minutes).

Then, the same children were taken into a rehabilitation program in which 16 sessions (8 weeks x 2 days a week) the HS device (30 minutes) and NDT (15 minutes) (HS + NDT method) were used together.

#### **Hippotherapy Simulator System Protocol**

HRS is a simulator consisting of a seat (saddle), control panel, foot pedals, and hand grip, and has four different speed programs (warm-up, level 1-2-3). HRS is a device that moves forward, backward, backward-to-back, right-to-left swing and up-and-down swing in 3 dimensions, similar to the movements of a real horse, forming an 8-shaped movement on five axes. After the children sat in the saddle section, they were first taken to the warm-up speed program for 5 minutes, then to another one of the other speed levels (gradually moved to other speed levels

as appropriate for the development and tolerance of children) and finally to the warm-up speed program for 5 minutes.

### Neurodevelopmental Therapy Based Rehabilitation

NDT rehabilitation program was determined according to the children's level of gross motor function, age, gender, mental state, and preferences.

NDT program consists of the rehabilitation of muscle tone disorders, increasing sensory-perception-motor integrity, exercises to increase limb functions and body control, stretching and strengthening exercises for muscle shortness and weakness, exercises that include movements in daily life and training activities such as standing, walking, body care.

Statistical Analysis Plan (SAP)

(Pages 7-8)

**January 11, 2018** 

#### **Statistical Analysis Plan (SAP)**

For the data analysis of our research, an 11.5 version of the statistical program "SPSS (Statistical Package for Social Science) for Windows" was used in the computer environment. With the statistical program, 95 percentage confidence interval and significance were evaluated at p < 0.05 level.

The conformity of the data to normal distribution was analyzed with the "Kolmogorov Smirnov" test. In the Kolmogorov Smirnov test, it was decided that the distributions did not conform to the normal distribution, since p < 0.05 and histogram graphics were skewed. For this reason, analyzes were performed using nonparametric statistical methods.

"Friedman Test (variance analysis in repetitive measurements)" was used to compare the evaluations made after the initial, NDT approach and after the HS + NDT method, and to compare the changes between the results obtained. The pairwise comparisons of the changes in the evaluation results obtained after the Friedman test were analyzed with the "Wilcoxon signed-rank test". Bonferonni correction was made after the Friedman test. As a result, the significance value of 0.05 was divided by 3 and the new significance value was determined as 0.016.

**Informed Consent Form (ICF)** 

(Pages 9 - 13)

**January 11, 2018** 

#### **Informed Consent Form (ICF)**

#### **Description of the Physiotherapist**

This study, which your child will participate in, is scientific research and is called "The Effects of a Hippotherapy Simulator in Children with Cerebral Palsy". This study aims to research the effect of simulated hippotherapy to correct problems related to standing and sitting balance, gait, trunk involvement, and functionality of your lower limbs in children with spastic cerebral palsy.

The research will be carried out by R.A Pt. Canan GÜNAY YAZICI (Tel: +90 538 460 12 49), under the supervision of Zübeyir SARI, Ph.D., Assoc. Prof. Dr., Marmara University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, as a master thesis at "The Private Dilbade Special Education and Rehabilitation Center".

If you agree to participate in the study, your child will be taken to a 16-week physiotherapy and rehabilitation program by physiotherapists. After socio-demographic information about you and your child is obtained before the treatment program, your child's gross motor functions, angle measurements of the lower extremity joints and muscle tone, gait analysis, trunk affection, balance, and daily functions will be evaluated. After the first evaluation, your child will be taken to the 8-week neurodevelopmental treatment program that is routinely applied. After this program is over, your child will be included in the hippotherapy simulator treatment that mimics the movements of a real horse in addition to the neurodevelopmental treatment program. Initial assessments will be repeated at the end of the 8th week and 16th week of the rehabilitation. Your responsibilities regarding this research are to pay attention to your sessions and to follow the suggestions. You should regularly attend a 45-minute session 2 days a week for this study, which is planned to last 16 weeks.

Your child is being invited to a research project. You need to understand why and how this research will be done before making a decision. Please take some time and read the following pieces of information carefully, discuss it with others if you wish. If you have an unclear section or need more detailed information, you can get information from us. You are invited to our research because we think your child matches the criteria to be included. We would like to note that participation is voluntary and that refusal to participate does not lead to any penalty or loss of any benefit. In the same way, you can withdraw from the research at any time.

All your medical and identification information about you and your child will be kept confidential and your identity information will not be provided even if the research is published, but the audience of the research, the attendants, ethical committees and government authorities can access your medical information when necessary. When you want, you can access medical information about yourself and your child.

The evaluation methods and treatment programs to be applied in our study have no known harm or risk. In this regard, you and your child can be safe and comfortable. In case of any unexpected damage during the evaluation and rehabilitation process, you will be informed immediately. In case of any damage to the participants, the necessary applications will be covered by the researchers without any resources. For this, you will not be charged any fees, neither you nor your social security insurance.

While participation in the research does not help you immediately, it is hoped that our research results will have benefits for the organization, society or science in the future. No fee will be charged for this study from you or the social security institution to which you are affiliated.

#### **Consent of the Participant**

I have read this entire written document. Since I don't know reading/language, it was understandably read and explained or translated to me. I was allowed to ask, evaluate and make decisions about my child's health status during and after my application and while filling out this form. All kinds of treatment, diagnosis, and alternatives including risks and dangers of treatment were explained. After all these explanations told to me and my child, I accept this invitation for scientific research with my consent.

| Name and the Surname of the Participant and Legal Representative: | |
|---|---|
| Date: | Signature: |
| Name and Surname of the Withness: | |
| Date: | Signature: |

#### **Declaration of the Physiotherapist**

I gave the patient the necessary information about the study and the procedures to be performed. I believe that the patient understood this information, asked me the questions that she/he wanted to ask, and accepted the process with her/his free will.

Researcher: Physiotherapist Canan GÜNAY YAZICI

**Address:** Marmara University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation - Başıbüyük Maltepe/Istanbul/TURKEY

Mobile Phone: +90 538 460 12 49 E-mail: cnngnyzc@gmail.com

Date: Signature:

#### **Declaration of the Participant / Legal Representative**

Ms. Canan GÜNAY YAZICI said that medical research would be conducted and explained the above information about this research to me. I know that my child is invited to this research as a participant. If I participate in this research, I believe that the confidentiality of my child's information will be handled with great care and respect during the research. During the conduct of the study, information was provided that my child's personal information would be carefully protected. I also know that this information will only be used for educational and scientific purposes. During the research, I can withdraw from work at any time without any reason (However, in this case, I am aware of the difficult situation that the researchers will cause if I do not report anything). I do not take any financial responsibility for the research costs. There will be no payment for me. I will not be exposed to any monetary burden in any health problem that may arise directly or indirectly during the research. When we encounter any health problems during the research; I know that I can call the physiotherapist Canan GÜNAY YAZICI on an hour from +90 538 460 120 49 (mobile) phone.

We did not experience any compulsive behavior to participate in the research. I know that if we refuse to participate, this will not harm our current treatment and our relationship with the physiotherapist.

I understood all the explanations made to me in detail. At the end of a certain thinking period, I decided that my child could participate in this research project as a participant. I voluntarily accept this invitation on behalf of my child.

**Voluntary Approval Form** 

I have read the text above which shows the information that should be given to the

volunteer before investigating. These were written and was explained verbally. With these

conditions, I agree to participate in this research without any pressure or compulsion on me and

my child.

A signed copy of this four-page form will be given to me.

Name and the Surname of the Participant and Legal Representative:

Date: Signature:

Name and Surname of the Withness (who have witnessed the process of receipt until

the end):

Date: Signature:

The researcher who made the explanations,

Researcher: Physiotherapist Canan GÜNAY YAZICI

Address: Marmara University, Institute of Health Sciences, Department of

Physiotherapy and Rehabilitation - Başıbüyük Maltepe/Istanbul/TURKEY

Mobile Phone: +90 538 460 12 49 E-mail: cnngnyzc@gmail.com

Date: Signature:

**Annex 1.** Marmara University Faculty of Medicine Clinical Researches Ethics Committee Approval (Approval made at the meeting on 02.09.2016 with approval number: 09.2016.478)



#### Marmara Üniversitesi Tıp Fakültesi Klinik Araştırmalar Etik Kurulu

| | PROTOKOL KODU | 09.2016.478 |
|---|---|---|
| BAŞVURU<br>BİLGİLERİ | PROJE ADI | Serbral Palsi'li Çocuklarda simüle Hippoterapi Eğitiminin<br>Etkinliği |
| | SORUMLU ARAŞTIRICI ÜNVANI/ADI | Doç. Dr. Zübeyir SARI |

| h | arih 02.09.2016 | | | | |
|---|---|---|---|---|---|
| , | ukarıda başvuru bilgileri ver<br>İlnarak incelenmiş ve gerçek<br>onrasında yapılacak her türli<br>nayının yenilenmesi gerekmek | ilen araştırma başvuru dosyası v<br>leştirilmesinde sakınca bulunmad<br>ü proje değişiklikleri (katılımcıla<br>ttedir. | e ilgili belgeler araştır<br>lığı için Kurulumuzca<br>r, başlık vb.) veya pro | manın gerekçe, amaç,<br>onaylanmasına oy bir<br>otokol değişikliklerinin | yaklaşım ve yöntemleri dikka<br>liği ile karar verilmiştir. On:<br>Etik Kurula bildirilerek pro |
| YELER | | | | | |
| Unvani / Adı / Soyadı | Uzmanlık Dalı | Kurumu / EK Üyeliği | Onaylanan Proje<br>ile İlişkisi | Toplantiya<br>katılım | ĺmza |
| Prof.Dr. Haner DİRESKENELİ | Romatoloji | M.Ü Tıp Fakültesi/ Başkan | Var Yok | Evet Hayır | 4 |
| Prof.Dr. Tülin ERGUN | Dermatoloji | M.Ü Tıp Fakültesi/Başkan<br>Yrd. | <br>Var Yok | Evet Hayır | \$ |
| Prof.Dr. Handan KAYA | Patoloji | M.Ü Tıp Fakültesi/Üye | <br>Var Yok | Evet Hayır | 4 |
| Prof.Dr. M.Bahadır GÜLLÜOĞ | LU Genel Cerrahi | M.Ü Tıp Fakültesi/Üye | Var Yok | Evet Hayır | hoping - |
| Prof.Dr. Atila KARAALP | Farmakoloji | M.Ü Tıp Fakültesi/Üye | Var Yok | EVET HAYIR | ATTH |
| Prof.Dr. Semra SARDAŞ | Eczacı | M.Û Eczacılık Fak/Üye | <br>Var Yok | Evet Hayır | Ma |
| Prof.Dr. Başak DOĞAN | Diş Hekimi | M.Ü Diş Hekimliği Fak./Üye | Var Yok | Evet Hayır | |
| Prof. Dr. Beste Melek ATASOY | Radyasyon<br>Onkolojisi | M.Û Tıp Fakültesi/Üye | · · · Var Yok | Evet Hayır | , |
| Doç. Dr. Elif KARAKOÇ AYDIN | Çocuk Sağlığı ve<br>Hastalıkları | M.Ü Tıp Fakültesi/Üye | · · · Var Yok | Evet Hayır | No. |
| Doç.Dr. Meltem KORAY | Diş Hekimi | İstanbul Üniv. Diş Hekimliği<br>Fak./Üye | Var Yok | Evet Hayır | <i></i> |
| Doç.Dr. Tolga GÜVEN | Tıp Tarihi ve Etik | M.Ü Tıp Fakültesi/Üye | · · · Var Yok | Evet Hayır | |
| Doç. Dr. Gürkan SERT | Hukukçu | M.Ü Tıp Fakültesi/Üye | · · · Var Yok | Evet Hayır | 8 |
| Yrd.Doç.Dr: Figen DEMİR | Halk Sağlığı | Acıbadem Üniv. Tıp Fak. | <br>Var Yok | Evet Hayır | A |
| Yrd.Doç.Dr. Pınar Mega TİBER | Biyofizik | M.Ü Tıp Fakültesi/Üye | · · · Var Yok | Evet Hayır | 10 |
| Gözde Aynur MİRZA | Sağlık Mensubu<br>olmayan kişi | Serbest | Var Yok | Evet Hayır | gyw |

# **Annex 2. Participants Tracking Form**

| No. | | Date. | | |
|----------------------|-------------|-----------|--------|------------|
| Name-Surname | | ' | | |
| Name-Sumame | | | | |
| Address | | | | |
| 7 Iddiess | | | | |
| Phone | | | | 1 |
| Gender | Female | Male | Age | |
| Height | | + | Weight | |
| CP Type | Hemiparesis | Diparesis | Quad | driparesis |
| GMFCS Level | I | II 🔲 | III | |
| Education Level | | | | |
| Having surgery/date | | | | |
| Botulinum toxin | | | | |
| injections./date | | | | |
| Auxiliary tool used | | | | |
| Orthotic/device used | | | | |

## PASSIVE RANGE OF MOTION

| MEASURE | BEFORE | | 8. WEEKS | | 16.WEEKS | |
|-----------------------|--------|-------|----------|-------|----------|-------|
| | LEFT | RİGHT | LEFT | RİGHT | LEFT | RİGHT |
| Hip flexion | | | | | | |
| Hip extension | | | | | | |
| Hip internal rotation | | | | | | |
| Hip external rotation | | | | | | |
| Hip abduction | | | | | | |
| Hip adduction | | | | | | |
| Knee flexion | | | | | | |
| Knee extension | | | | | | |
| Dorsiflexion | | | | | | |
| Plantar flexion | | | | | | |
| Trunk lateral flexion | | | | | | |
| Trunk flexion | | | | | | |
| Trunk extension | | | | | | |

### MODIFIED ASHWORTH SCALE

| MEASURE | BEFORE | | 8. WEEKS | 16.WEEKS | |
|---------------|--------|-------|----------|----------|-------|
| | LEFT | RİGHT | LEFT | LEFT | RİGHT |
| Hip flexion | | | | | |
| Hip abduction | | | | | |
| Hamstring | | | | | |
| Quadriceps | | | | | |
| Gastrocnemius | | | | | |
| Soleus | | | | | |

| Grade | Description |
|---|---|
| 0 | No increase in muscle tone |
| 1 | Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part/s is/are moved in flexion or extension. |
| 1+ | Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM. |
| 2 | More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved. |
| 3 | Considerable increase in muscle tone, passive movement difficult. |
| 4 | Affected part(s) rigid in flexion or extension. |

ROM, range of motion.

## MYOTON®PRO DIGITAL PALPATION DEVICE

| MEASURE | BEFORE | | 8. WEEKS | 16.WEEKS | |
|---|---|---|---|---|---|
| | LEFT | RİGHT | LEFT | LEFT | RİGHT |
| Hip flexion | | | | | |
| Hip adduction | | | | | |
| Hamstring (semitendinosus, biceps femoris) | | | | | |
| Quadriceps (rectus<br>femoris, vastus lateralis,<br>vastus medialis) | | | | | |
| Gastrocnemius | | | | | |
| Soleus | | | | | |

## GROSS MOTOR FUNCTIONAL CLASSIFICATION SYSTEM (GMFCS)

## Level of the participant:



### THE TRUNK IMPAIRMENT SCALE

| Iten | 1 | | |
|---|---|---|---|
| 1 | Static sitting balance<br>Starting position | Patient falls or cannot maintain starting position for 10 seconds without arm support Patient can maintain starting position for 10 seconds If score = 0, then TIS total score = 0 | □ 0<br>□ 2 |
| 2 | Starting position Therapist crosses the unaffected leg over the hemiplegic leg | Patient falls or cannot maintain sitting position for 10 seconds without arm support Patient can maintain sitting position for 10 seconds | □ 0<br>□ 2 |
| 3 | Starting position Patient crosses the unaffected leg over the hemiplegic leg | Patient falls Patient cannot cross the legs without arm support on bed or table Patient crosses the legs but displaces the trunk more than 10 cm backwards or assists crossing with the hand Patient crosses the legs without trunk displacement or assistance Total static sitting balance | □ 0<br>□ 1<br>□ 2<br>□ 3 |
| | Dynamic sitting balance Starting position Patient is instructed to touch the bed or table with the hemiples elbow (by shortening the hemiplegic side and lengthening the unaffected side) and return to the starting position | Patient falls, needs support from an upper extremity or the elbow ic does not touch the bed or table Patient moves actively without help, elbow touches bed or table If score = 0, then items 2 and 3 score 0 | □ 0<br>□ 1 |
| | 2 Repeat item 1 | Patient demonstrates no or opposite shortening/lengthening Patient demonstrates appropriate shortening/lengthening If score = 0, then item 3 scores 0 | □ 0<br>□ 1 |
| | 3 Repeat item 1 | Patient compensates. Possible compensations are: (1) use of upper extremity, (2) contralateral hip abduction, (3) hip flexion (if elbow touches bed or table further then proximal half of femur), (4) knee flexion, (5) sliding of the feet Patient moves without compensation | □ 0<br>□ 1 |
| | 4 Starting position Patient is instructed to touch the bed or table with the unaffect elbow (by shortening the unaffected side and lengthening the hemiplegic side) and return to the starting position | Patient falls, needs support from an upper extremity or the elbow does not touch the bed or table Patient moves actively without help, elbow touches bed or table If score = 0, then items 5 and 6 score 0 | □ 0<br>□ 1 |
| | 5 Repeat item 4 | Patient demonstrates no or opposite shortening/lengthening Patient demonstrates appropriate shortening/lengthening If score = 0, then item 6 scores 0 | □ 0<br>□ 1 |

| ( | 6 | Repeat item 4 | Patient compensates. Possible compensations are: (1) use of upper extremity, (2) contralateral hip abduction, (3) hip flexion (if elbow touches bed or table further then proximal half of femur) (4) knee flexion, (5) sliding of the feet Patient moves without compensation | |
|---|---|---|---|---|
| | 7 | Starting position Patient is instructed to lift pelvis from bed or table at the hemiplegic side (by shortening the hemiplegic side and lengthening the unaffected side) and return to the starting position | Patient demonstrates no or opposite shortening/lengthening g Patient demonstrates appropriate shortening/lengthening If score = 0, then item 8 scores 0 | □ (<br>□ 1 |
| { | 3 | Repeat item 7 | Patient compensates. Possible compensations are: (1) use of upper extremity, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation | |
| Ċ | ) | Starting position Patient is instructed to lift pelvis from bed or table at the unaffected side (by shortening the unaffected side and lengthening the hemiplegic side) and return to the starting position | Patient demonstrates no or opposite shortening/lengthening Patient demonstrates appropriate shortening/lengthening If score = 0, then item 10 scores 0 | □ (<br>□ 1 |
| 1 | 10 | Repeat item 9 | Patient compensates. Possible compensations are: (1) use of upper extremities, (2) pushing off with the ipsilateral foot (heel loses contact with the floor) Patient moves without compensation Total dynamic sitting balance | □ (<br>□ 1<br>/1( |
| 1 | S<br>P<br>sh | Co-ordination tarting position atient is instructed to rotate upper trunk 6 times (every shoulder nould be moved forward 3 times), first side that moves must be emiplegic side, head should be fixated in starting position | Rotation is asymmetrical Rotation is symmetrical If score = 0, then item 2 scores 0 | □ 0<br>□ 1<br>□ 2 |
| 2 | R | epeat item 1 within 6 seconds | • | □ 0<br>□ 1 |
| 3 | P<br>sł | tarting position<br>atient is instructed to rotate lower trunk 6 times (every knee<br>nould be moved forward 3 times), first side that moves must be<br>emiplegic side, upper trunk should be fixated in starting position | Rotation is asymmetrical | □ 0<br>□ 1<br>□ 2 |
| 4 | R | epeat item 3 within 6 seconds | | □ 0<br>□ 1<br>/6 |
| | | | Total Trunk Impairment Scale | /23 |

#### PEDIATRIC BALANCE TEST

All items are scored between 0 and 4 and the total score is calculated.

| | Pediatric Balance Scale Items |
|----|----------------------------------------|
| 1 | Sitting to standing |
| 2 | Standing to sitting |
| 3 | Transfers |
| 4 | Standing unsupported |
| 5 | Sitting unsupported |
| 6 | Standing with eyes closed |
| 7 | Standing with feet together |
| 8 | Standing with one foot in front |
| 9 | Standing on one foot |
| 10 | Turning 360 degrees |
| 11 | Turning to look behind |
| 12 | Retrieving object from floor |
| 13 | Placing alternate foot on stool |
| 14 | Reaching forward with outstretched arm |

## THE FUNCTIONAL INDEPENDENCE MEASURE (WEEFIM) (WEE-FIM)

| Items | Descriptive Items |
|---------------------------------------|--------------------|
| Domain 1: self-care | |
| (maximum = 56) | |
| 1 | Eating |
| 2 | Grooming |
| 2 3 | Bathing |
| 4 5 | Dressing-upper |
| 5 | Dressing-lower |
| 6 | Toileting |
| 7 | Bladder |
| 8 | Bowel |
| Domain 2: mobility | |
| (maximum = 35) | |
| 9 | Chair transfer |
| 10 | Toilet transfer |
| 11 | Tub transfer |
| 12 | Walk |
| 13 | Stairs |
| Domain 3: cognition<br>(maximum = 35) | |
| 14 | Comprehension |
| 15 | Expression |
| 16 | Social interaction |
| 17 | Problem solving |
| 18 | Memory |
| Total scores = 126 | |

| 7 = Fully independent<br>6 = Modified independent | Unaided |
|---|---|
| 5 = Surveillance is required<br>4 = Minimal aid (75% of children)<br>3 = Moderate help (50% of children) | Helped / Modified Dependent |
| 2 = Maximum help (25% of children)<br>1 = Full help ( <less 25%="" children="" do)<="" of="" td="" than=""><td>Totally Dependent</td></less> | Totally Dependent |

### **GROSS MOTOR FUNCTION MEASURE-88**

| Ite | m | A: LYING & ROLLING | _ | SCOR | Ę | _ | NT |
|---|---|---|---|---|---|---|---|
| | 1. | SUP, HEAD IN MIDLINE: TURNS HEAD WITH EXTREMITIES SYMMETRICAL | 0 | 10 | 2□ | 3□ | 1. |
| * | 2. | SUP: BRINGS HANDS TO MIDLINE, FINGERS ONE WITH THE OTHER | 0 | 1□ | 2□ | 3□ | 2. |
| | 3. | SUP: LIFTS HEAD 45° | 0 | 1 | 2□ | 3□ | 3. |
| | 4. | SUP: FLEXES R HIP & KINEE THROUGH FULL RANGE | 0 | 1 | 2□ | 3□ | 4. |
| | 5. | SUP: FLEXES L HIP & KNEE THROUGH FULL RANGE | 0 | 1□ | 2□ | 3□ | 5. |
| ± | 6. | SUP: REACHES OUT WITH R ARM, HAND CROSSES MIDLINE TOWARD TOY | 0 | 1 | 2□ | 3□ | 6. |
| ± | 7. | SUP: REACHES OUT WITH L ARM, HAND CROSSES MIDLINE TOWARD TOY | 0 | 1 | 2□ | 3□ | 7. |
| | 8. | SUP: ROLLS TO PR OVER R SIDE | 0 | 10 | 2□ | 3□ | 8. |
| | 9. | SUP: ROLLS TO PR OVER L SIDE | 0 | 1 | 2□ | 3□ | 9. |
| ± | 10. | PR: LFTS HEAD UPRIGHT | 0 | 10 | 2□ | 3□ | 10. |
| | 11. | PR ON FOREARMS: LIFTS HEAD UPRIGHT, ELBOWS EXT., CHEST RAISED | 0 | 10 | 2□ | 3□ | 11. |
| | 12. | PR ON FOREARMS: WEIGHT ON R FOREARM, FULLY EXTENDS OPPOSITE ARM FORWARD | 0 | 10 | 2□ | 3□ | 12. |
| | 13. | PR ON FOREARMS: WEIGHT ON L FOREARM, FULLY EXTENDS OPPOSITE ARM FORWARD | 0 | 10 | 2□ | 3□ | 13. |
| | 14. | PR: ROLLS TO SUP OVER R SIDE | 0 | 10 | 2 | 3□ | 14. |
| | 15. | PR: ROLLS TO SUP OVER L SIDE | 0 | 10 | 2 | 3□ | 15. |
| | 16. | PR: prvots to R 90° using extremities | 0 | 10 | 2 | 3□ | 16. |
| | 17. | PR: PIVOTS TO L 90° USING EXTREMITIES | | 10 | 20 | 3□ | 17. |
| | | TOTAL DIMENSION A | | | | | |
| lte: | | B: SITTING | | SCOR | - | | NT |
| • | 18. | SUP, HANDS GRASPED BY EXAMINER: PULLS SELF TO SITTING WITH HEAD CONTROL | U— | 10 | 2 | 3□ | 18. |
| | 19. | SUP: ROLLS TO R SIDE, ATTAINS SITTING | - | 10 | 2 | 3□ | 19. |
| | 20. | SUP: ROLLS TO L SIDE, ATTAINS SITTING | 0 | 1 | 2 | 3□ | 20. |
| * | 21. | SIT ON MAT, SUPPORTED AT THORAX BY THERAPIST: LIFTS HEAD UPRIGHT, MAINTAINS 3 SECONDS | 0 | 1 | 2□ | 3□ | 21. |
| • | 22. | SIT ON MAT, SUPPORTED AT THORAX BY THERAPIST: LIFTS HEAD MIDLINE, MAINTAINS 10 SECONDS | 0□ | 1□ | 2 | 3□ | 22. |
| ± | 23. | SIT ON MAT, ARM(S) PROPPING: MAINTAINS, 5 SECONDS | 0 | 10 | 2□ | 3□ | 23. |
| * | 24. | SIT ON MAT: MAINTAIN, ARMS FREE, 3 SECONDS | _ | 1□ | 2□ | 3□ | 24. |
| * | 25. | SIT ON MAT WITH SMALL TOY IN FRONT: LEANS FORWARD, TOUCHESTOY, RE-ERECTS WITHOUT ARM PROPPING | 0 | 1 | 2□ | 3□ | 25. |
| ± | 26. | SIT ON MAT: TOUCHES TOY PLACED 45° BEHIND CHILD'S R SIDE, RETURNS TO START | 0 | 1□ | 2□ | 3□ | 26. |
| ± | 27. | SIT ON MAT: TOUCHES TOY PLACED 45° BEHIND CHILD'S L SIDE, RETURNS TO START | 0 | 10 | 2 | 3□ | 27. |
| | 28. | R SIDE SIT: MAINTAINS, ARMS FREE, 5 SECONDS | 0□ | 10 | 2 | 3□ | 28. |
| | 29. | L SIDE SIT: MAINTAINS, ARMS FREE, 5 SECONDS | 0 | 10 | 2 | 3□ | 29. |
| ± | 30. | SIT ON MAT: LOWERS TO PR WITH CONTROL | 0 | 10 | 2 | 3□ | 30. |
| * | 31. | SIT ON MAT WITH FEET IN FRONT: ATTAINS 4 POINT OVER R SIDE | 0 | 10 | 2□ | 3□ | 31. |
| * | 32. | SIT ON MAT WITH FEET IN FRONT: ATTAINS 4 POINT OVER L SIDE | • | 10 | 2□ | 3□ | 32. |
| | 33. | SIT ON MAT: PIVOTS 90°, WITHOUT ARMS ASSISTING | - | 10 | 2□ | 3□ | 33. |
| ± | 34. | SIT ON BENCH: MAINTAINS, ARMS AND FEET FREE, 10 SECONDS | _ | 10 | 2 | 3□ | 34. |
| ± | 35. | STD: ATTAINS SIT ON SMALL BENCH | - | 10 | 2 | 3□ | 35. |
| ± | 36. | ON THE FLOOR: ATTAINS SIT ON SMALL BENCH | _ | 10 | 20 | 3□ | 36. |
| * | 37. | ON THE FLOOR: ATTAINS SIT ON LARGE BENCH | - | 10 | 2□ | 3□ | 37. |
| | | | _ | ,_ | | | |
| | | TOTAL DIMENSION B | | | | | |

| Ite | m | C: CRAWLING & KNEELING | _ | SC | ORE | | NT |
|---|---|---|---|---|---|---|---|
| | 38. | PR: creeps forward 1.8m (6') | 0 | 10 | 2 | 3□ | 38. |
| * | 39. | 4 POINT: MAINTAINS, WEIGHT ON HANDS AND KNEES, 10 SECONDS | 0 | 1 | $_2\square$ | 3□ | 39. |
| * | 40. | 4 POINT: ATTAINS SIT ARMS FREE | 0 | 1 | $_2\square$ | 3□ | 40. |
| * | 41. | PR: ATTAINS 4 POINT, WEIGHT ON HANDS AND KNEES | 0 | 1 | $_2\square$ | 3□ | 41. |
| * | 42. | 4 POINT: REACHES FORWARD WITH R ARM, HAND ABOVE SHOULDER LEVEL | 0 | 1□ | $_2\square$ | 3□ | 42. |
| * | 43. | . 4 POINT: REACHES FORWARD WITH L ARM, HAND ABOVE SHOULDER LEVEL | | 43. | | | |
| * | 44. | 4 POINT: crawls or hitches forward 1.8m(6') | 0 | 1 | $_2\square$ | 3□ | 44. |
| * | 45. | 4 POINT: crawLs reciprocally forward 1.8m ( 6') | 0 | 1 | $_{2}\square$ | 3□ | 45. |
| * | 46. | 4 POINT: CRAWLS UP 4 STEPS ON HANDS AND KNEES/FEET | 0 | 1 | $_{2}\square$ | 3□ | 46. |
| | 47. | 4 POINT: CRAWLS BACKWARDS DOWN 4 STEPS ON HANDS AND KNEES/FEET | 0 | 1 | 2□ | 3□ | 47. |
| * | 48. | SIT ON MAT: ATTAINS HIGH KN USING ARMS, MAINTAINS, ARMS FREE, 10 SECONDS | 0 | 1 | $_{2}\square$ | 3□ | 48. |
| | 49. | HIGH KN: ATTAINS HALF KN ON R KNEE USING ARMS, MAINTAINS, ARMS FREE, 10 SECONDS | 0 | 1 | 2 | 3□ | 49. |
| | 50. | HIGH KN: ATTAINS HALF KN ON L KNEE USING ARMS, MAINTAINS, ARMS FREE, 10 SECONDS | | 1 | $_{2}\square$ | 3□ | 50. |
| * | 51. | HIGH KN: KN WALKS FORWARD 10 STEPS, ARMS FREE | 0 | 1 | 2 | 3□ | 51. |
| | | TOTAL DIMENSION C | | | | | |

| Ite | m | D: STANDING | | SC | DRE | | NT |
|---|---|---|---|---|---|---|---|
| * | 52. | ON THE FLOOR: PULLS TO STD AT LARGE BENCH | 0 🗆 | 10 | 2 | 3□ | 52. |
| * | 53. | STD: MAINTAINS, ARMS FREE, 3 SECONDS | 0 | 1 | $_{2}\square$ | 3□ | 53. |
| * | 54. | STD: HOLDING ON TO LARGE BENCH WITH ONE HAND, LIFTS R FOOT, 3 SECONDS | 0 | 1 | 2 | 3□ | 54. |
| * | 55. | STD: HOLDING ON TO LARGE BENCH WITH ONE HAND, LIFTS L FOOT, 3 SECONDS | 0 | 1 | 2 | 3□ | 55. |
| * | 56. | STD: maintains, arms free, 20 seconds | 0 | 1 | 2 | 3□ | 56. |
| * | 57. | STD: ufts L foot, arms free, 10 seconds | 0 | 1 | 2 | 3□ | 57. |
| * | 58. | STD: ufts R foot, arms free, 10 seconds | 0 | 1 | 2 | 3□ | 58. |
| * | 59. | SIT ON SMALL BENCH: ATTAINS 5TD WITHOUT USING ARMS | 0 | 1 | 2 | 3□ | 59. |
| * | 60. | HIGH KN: ATTAINS STD THROUGH HALF KN ON R KNEE, WITHOUT USING ARMS | 0 | 1 | 2 | 3□ | 60. |
| * | 61. | HIGH KN: ATTAINS STD THROUGH HALF KN ON L KNEE, WITHOUT USING ARMS | 0 | 1 | 2 | 3□ | 61. |
| * | 62. | STD: LOWERS TO SIT ON FLOOR WITH CONTROL, ARMS FREE | 0 | 1 | 2 | 3□ | 62. |
| * | 63. | STD: ATTAINS SQUAT, ARMS FREE | 0 | 1 | 2 | 3□ | 63. |
| * | 64. | STD: PICKS UP OBJECT FROM FLOOR, ARMS FREE, RETURNS TO STAND | 0 | 1 | 2 | 3□ | 64. |
| | | TOTAL DIMENSION D | | | | | |

| Item | | E: WALKING, RUNNING & JUMPING | | SCOR | | • | NT |
|---|---|---|---|---|---|---|---|
| * | 65. | STD, 2 HANDS ON LARGE BENCH: cruises 5 steps to R | 0 | 10 | 2 | 3 | 65. |
| * | 66. | STD, 2 HANDS ON LARGE BENCH: cruises 5 steps to L | 0 🗆 | 1 u | 2 | 3□ | 66. |
| * | 67 | STD, 2 HANDS HELD: WALKS FORWARD 10 STEPS | 0 🗆 | 1 | 2 | 3□ | 67. |
| * | 68. | STD, 1 HAND HELD: walks forward 10 steps | 0 🗆 | 1 | 2 | 3□ | 68. |
| * | 69. | STD: walks forward 10 steps | 0 🗆 | 1 🗆 | 2 | 3□ | 69. |
| * | 70. | STD: walks forward 10 steps, stops, turns 180°, returns | 0 🗆 | 1 | 2 | 3□<br>3□ | 70. |
| * | 71 | STD: WALKS BACKWARD 10 STEPS | 0 🗆 | 1 | 2 | 3□ | 71. |
| * | 72. | STD: WALKS FORWARD 10 STEPS, CARRYING A LARGE OBJECT WITH 2 HANDS | 0 🗆 | 1 | 2 | 3□ | 72. |
| * | 73 | STD: walks forward 10 consecutive steps between parallel lines 20cm (8")apart | 0 🗆 | 10 | 2 | 3□<br>3□ | 73. |
| * | 74. | STD: WALKS FORWARD 10 CONSECUTIVE STEPS ON A STRAIGHT LINE 2cm (3/4") WIDE | 0 🗆 | 10 | 2 | 3<br>3 | 74. |
| * | 75. | STD: STEPS OVER STICK AT KNEE LEVEL, R FOOT LEADING | 0 🗆 | 10 | 2 | 3<br>3 | 75. |
| * | 76. | STD: STEPS OVER STICK AT KNEE LEVEL, L FOOT LEADING | o□ | 1<br>1 | 2□ | 3□ | 76. |
| * | 77. | STD: runs 4.5m (15'), stops & returns | n 🗆 | 10 | 2□ | 3□ | 77. |
| * | <b>7</b> 8. | STD: KICKS BALL WITH R FOOT | n□ | 10 | 2 | 3 | <b>78</b> . |
| * | <b>7</b> 9. | STD: KICKS BALL WITH L FOOT | n□ | 1 | 2 | 3<br>3 | <b>7</b> 9. |
| * | 80. | STD: JUMPS 30cm (12") HIGH, BOTH FEET SIMULTANEOUSLY | 0 🗆 | 10 | 2 | 3□ | 80. |
| * | 81. | STD: Jumps forward 30 cm (12"), both feet simultaneously | 0 🗆 | 1 | 2 | 3□ | 81. |
| * | 82. | STD ON R FOOT: HOPS ON R FOOT 10 TIMES WITHIN A 60cm (24") CIRCLE | n 🗆 | 1 | 2 | 3 | 82. |
| * | 83. | STD ON L FOOT: HOPS ON L FOOT 10 TIMES WITHIN A 60cm (24") CIRCLE | 0 | 1□ | 2 | 3□ | 83. |
| * | 84. | STD, HOLDING 1 RAIL: WALKS UP 4 STEPS, HOLDING 1 RAIL, ALTERNATING FEET | ٥ | 1□ | 2 | 3□ | 84. |
| * | 85. | STD, HOLDING 1 RAIL: WALKS DOWN 4 STEPS, HOLDING 1 RAIL, ALTERNATING FEET | 0 | 1 | 2 | 3□ | 85. |
| * | 86. | STD: WALKS UP 4 STEPS, ALTERNATING FEET | 0 | 1□ | 2 | 3□ | 86. |
| * | 87. | STD: WALKS DOWN 4 STEPS, ALTERNATING FEET | 0 | 1□ | 2 | 3□ | 87. |
| * | 88. | STD ON 15cm (6") STEP: JUMPS OFF, BOTH FEET SIMULTANEOUSLY | • | 1□ | 2 | 3□ | 88. |
| | | | | | _ | - | |

| TOTAL DIMENSION E |
|-------------------|